CLINICAL TRIAL: NCT01180868
Title: The Biodistribution of 1-L-(2 Deoxy-2,- 18 Fluoroarabinofuranosyl) Cytosine ([18F]L-FAC) in Healthy Subjects and Patients With Cancer, Autoimmune and Inflammatory Diseases
Status: Completed | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-02-049; DE-PS02-08ER08-01 (Other Grant/Funding Number: Department of Energy); CIRM No. RT1-01126-1 (Other Grant/Funding Number: California Institute for Regenerative Medicine)
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Autoimmune Diseases; Cancer
Keywords: imaging probe; cancer; inflammatory tissue; inflammatory diseases
MeSH Terms: conditions — Autoimmune Diseases; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- patients with cancer: patients with hematological malignancies and solid tumors
- patients with autoimmune dosorders: patients with Rheumatoid arthritis, Crohns's disease, systemic lupus erythematosus.
- healthy subjects

SUMMARY:
The purpose of this study is to determine the biodistribution of a new agent 1-L-(2 deoxy-2,-18fluoroarabinofuranosyl) cytosine non-invasively in healthy humans and to evaluate whether it can be used to image cancer, autoimmune disease, and inflammation

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years of age
* women of childbearing potential will undergo a pregnancy test free of charge
* patients with hematological malignancies, solid tumors or autoimmune disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with cancer, patients with autoimmune dosorders, and healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-05; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Schiepers, M.D. Ph.D, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States